CLINICAL TRIAL: NCT02027129
Title: Comparison of Cardio-respiratory Variables Between Low-frequency High Frequency Oscillation With/Without Tracheal Gas Insufflation and High-frequency High-frequency Oscillation in Severe ARDS.
Brief Title: Physiological Study of Low-frequency HFO/HFO-TGI and High-frequency HFO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Spyros D. Mentzelopoulos, Assistant Professor in Intensive Care Medicine, University of Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 271-30-10-2013
Record Dates: First submitted 2014-01-02; First posted 2014-01-03 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Cor Pulmonale
Keywords: Respiratory Distress Syndrome, Adult; Cor Pulmonale; High Frequency Ventilaiton
MeSH Terms: conditions — Respiratory Distress Syndrome; Pulmonary Heart Disease | interventions — High-Frequency Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low frequency HFO/HFO-TGI vs high frequency HFO (Other): Total study population for the testing of the ventilatory strategies
  Interventions: Other: High Frequency Oscillation

INTERVENTIONS:
Other: High Frequency Oscillation — Comparison of low frequency HFO/HFO-TGI with cuff leak and high frequency HFO without cuff leak on right ventricular function

SUMMARY:
Recent data from large trials of high-frequency high frequency oscillation (HFO) without a cuff leak vs, lung-protective conventional ventialtion (CMV) failed to show any HFO-related benefit with respect to outcome. A possible explanation is that HFO increases the probability of right ventricular dysfunction due to the combination of high mean airway pressures (mPaws) and hypercapnia. In contrast, available preliminary data on low-frequency HFO-tracheal gas insufflation (TGI) with cuff leak vs. CMV are suggestive of an HFO-TGI related benefit. Low-frequency HFO-TGI with a cuff leak is associated with relatively low mean tracheal pressures and adequate control of PaCO2. Thus, the investigators intend to test the hypothesis that low frequency HFO +/- TGI with a cuff leak is associated with better right ventricular function relative to high-frequency HFO without a cuff leak.

DETAILED DESCRIPTION:
Rationale of the study Acute Respiratory Distress Syndrome (ARDS) is an acute inflammatory state of the pulmonary parenchyma that causes hypoxemia, atelectasis, pulmonary congestion, and reduction in pulmonary compliance. Mechanical ventilation is actually life-saving, but it may traumatize the lungs (e.g. volutrauma, barotrauma, atelectrauma, and biotrauma). The use of low tidal volumes and high positive end-expiratory pressure (PEEP), aims at attenuating ventilator-associated lung injury. However, ARDS mortality still remains high. High frequency oscillation (HFO) is an alternative ventilatory technique that employs very low tidal volumes (1-4 ml/kg) administered at high frequencies (3-15 Hz). Prior observational studies have reported improvements in oxygenation, whereas recent two-center data on severe ARDS suggest a survival benefit from the intermittent, combined use of low-frequency HFO with a cuff leak, Recruitment maneuvers (RMs), and tracheal gas insufflation (TGI). The addition of TGI improves oxygenation and CO2 elimination; however, it is still unclear whether it affects survival. Two recently published multicenter studies showed either neutral (10) or negative results (11) with respect to survival when high frequency HFO without a cuff leak was used in the treatment of early ARDS. However, these negative results may be partly due to right ventricular overload/dysfunction/failure caused by the combination of high intrathoracic pressures and hypercapnia, with consequent hemodynamic instability and increased need of inotropic/vasopressor support. Accordingly, the investigators hypothesize that a different HFO strategy [employing a combination of a low frequency and a cuff leak - which augments CO2 elimination and is associated with relatively low mean tracheal pressures - could lead to different results.

A high intrathoracic pressure may impede venous return and increase pulmonary vascular resistance. This concurrent right ventricular preload reduction and afterload increase might cause right ventricular dysfunction/failure. On the other hand, the placement of a cuff leak results in a lower (by approx. 5-6 cmH2O) mean tracheal pressure relative to the set HFO-ventilator mean airway pressure (mPaw), with consequent unloading of the right ventricle. In addition, further unloading of the right ventricle can be expected through the combined use of a cuff leak, TGI, and a high HFO bias flow; these measures improve PaCO2 control and may prevent excessive, hypercapnia-induced increases in pulmonary vascular resistance. Right ventricular function can be assessed by transesophageal echocardiography (TEE) as previously described. Right ventricular dysfunction and associated dilatation may cause cardiac output reduction and coronary hypoperfusion; the latter may further compromise right ventricular performance and contribute to right ventricular failure.

The main goal of the present study is to document and compare the effect of lung protective conventional mechanical ventilation (CMV) and of different HFO strategies (already clinically tested in trials with conflicting results) on right ventricular performance as determined by TEE. More specifically, we intend to compare high-PEEP, lung protective CMV with a "high" mPaw/no cuff leak, high-frequency HFO strategy, and a "high" mPaw with cuff leak, "low" frequency HFO strategy with and without TGI.

Methods METHODS Eligible patients (relevant criteria provided below) with early and severe ARDS will be enrolled after the obtainment of informed, written, next-of-kin consent, as well as attending physician's non-written consent..

Patient monitoring will include electrocardiographic lead II, intra-arterial pressure (+/- cardiac index with PICCO plus, Pulsion Medical Systems, Munich, Germany)], and peripheral oxygen saturation (SaO2). Anesthesia will be maintained with midazolam and/or propofol, and fentanyl or remifentanil. Nrutomuscular blockade will be accomplished with cisatracurium, which will be used in concordance with current recommendations and as part of the attending physician-prescribed medical treatment. During the study period, all patients will be receiving a continuous infusion of cisatracurium.

CMV strategy Eligible study participants will have received at least 60 min of lung protective CMV with the following combinations of FiO2/PEEP: 0.5/10-12 cm H2O, 0.6/14-16 cm H2O, 0.7/14-16 cm H2O, 0.8/14-16 cm H2O, 0.9/16-18 cm H2O, 1.0/20-24 cmH2O. These combinations constitute "general" recommendations and further PEEP titrations of =< 4 cm H2O by attending physicians to the "best" combination of the patients' gas exchange and hemodynamic will be considered as acceptable. A high-PEEP-associated survival benefit has been recently documented. Whenever oxygenation deteriorates, PEEP will be increased first, followed by an increase in FiO2, while targeting "concordance" with the aforementioned FiO2/PEEP combinations.

Tidal volume will be within 5.5-7.5 mL/Kg predicted body weight. The maximal plateau pressure limit will be 40 cmH2O, and target plateau pressure will be ≤32 cmH2O; rationale: as in the study of Meade et al , a higher plateau pressure will be tolerated to allow for the use of a higher PEEP level. When plateau pressure exceeds 32 cmH2O for >15 min, the following adjustments will be conducted: tidal volume reduction up to 4.0 mL/kg predicted body weight, respiratory rate increase up to 35/min, and PEEP reduction by ≥2 cmH2O. These adjustments will have to concurrently result in the achievement of the below-provided gas-exchange targets.

The respiratory rate will be titrated to a pHa of 7.20-7.45. The inspiratory-to-expiratory time (Ι:Ε) ratio will be ≤1/2. The oxygenation target will be SaO2=90-95%, and/or PaO2=60-80 mmHg. At pHa<7.20, breathing circuit deadspace will be minimized by replacing the routinely used catheter mount by a short, low-volume angular connector, the tidal volume will be increased up to 8.0 mL/kg predicted body weight, and respiratory rate will be increased up to 35/min. If these measures fail, the criterion of "poor control of pHa/PaCO2," and the use of a bicarbonate infusion will be permitted. An additional option will be extracorporeal CO2 removal.

Algorithm of RMs and PEEP/FiO2

1. RM - Continuous positive airway pressure of 40-45 cmH2O for 40 sec, at an FiO2 of 1.0) and titration of PEEP and FiO2 so that SaO2=90-95%, or PaO2=60-80 mmHg (RMs may be repeated twice daily, once every 5 hours)
2. Reduction in FiO2 always precedes reduction in PEEP.
3. At FiO2=0.5 and PEEP<8 cmH2O - Weaning trial.
4. RMs may be administered for up to 5 days following the onset of the ARDS

HFO-RMs strategy

Previously published recommendations regarding HFO use (Sensormedics 3100B ventilator, Sensormedics, Yorba Linda, CA, USA) include the following steps:

1. Sufficient level of deep sedation/anesthesia for the abolishment of respiratory muscles activity, with or without neuromuscular blockade, so that patient-ventilator dyssynchrony is avoided.
2. Confirmation of endotracheal tube patency and placement of the tube at 3-4 cm above carina.
3. RMs: immediately after patient-oscillator connection, an RM will be performed (increase in the circuit pressure to 45 cmH2O for 40 sec with the oscillator's piston off). The RMs will be repeated just prior to changes in HFO frequency or just prior to/just after the initiation/termination of TGI.
4. FiO2 will initially be set at 1.0 and then reduced (over 10-15 min) to the FiO2 of the preceding CMV, provided that SaO2 is maintained >90%.
5. Bias flow will be set at 60 L/min to improve CO2 clearance from the breathing circuit.
6. I:E ratio will be maintained at 1:2.
7. According to the methods and results of preceding studies of the investigators, TGI will be equal to 50% of the preceding CMV minute ventilation.
8. The initial HFO mPaw will exceed the mPaw of the preceding CΜV by 8-10 cm H2O and will be titrated (by ±3 cmH2O) to the best oxygenation response (predicted to correspond to a "target" SaO2 of >= 95%) during a 60-min period of standard, low frequency HFO with cuff leak. The aforementioned period will precede the below-described 180-min period of HFO strategy testing.
9. Initial oscillation frequency will be randomly set at either at 3.5-4 Hz or at 7 Hz. The low frequency setting will be combined with a 3-5 cmH2O cuff leak and TGI for 60 min followed by "no-TGI" for another 60 min in random order. The high frequency setting will not be combined with either a cuff leak or TGI and will be maintained for an additional 60 min. Oscillatory pressure amplitude (ΔP) will be set at 90 cmH2O.

TEE measurements

The following parameters will be determined during baseline CMV:

Right ventricular diastolic area, left ventricular diastolic area, and Eccentricity Index. Assessment of coronary blood flow in the right main coronary artery and the left anterior descendant branch of the left main coronary artery (Note: coronary artery blood flow measurements proved technically difficult and time-consuming and were thus removed from the study protocol). The same measurements will be repeated at 120, 180, and 240 min after HFO initiation, and at 60 min following return to CMV. At the same time points, we will determine gas exchange, and hemodynamics including cardiac output with PICCO plus. Lastly, respiratory mechanics will be assessed with rapid end-expiratory/end-inspiratory airway occlusion during CMV.

Rescue oxygenation Rescue oxygenation methodology may include low-frequency HFO-TGI with cuff leak, prone positioning, inhaled nitric oxide, and extracorporeal membrane oxygenation. The duration of a rescue oxygenation session will be at least 10 hours with allowance for an unlimited extension if PaO2<60 mmHg. Rescue initiation criterion: PaO2<60 mmHg for more than 30 min at FiO2=1.0 during the high-PEEP, lung protective CMV, in the absence of any reversible cardio-respiratory pathology and/or ventilator malfunction.

Patient follow up Physiological variables (hemodynamics gas-exchange, and respiratory mechanics) and medication will be recorded within 2 hours before study enrollment and at 9 a.m. of days 1-10 following study enrollment. Organ dysfunction according to the Sequential Organ Dysfunction Assessment score and clinical course complications will be documented until day 60 post-enrollment. Lastly, the final outcome (i.e. survival to hospital discharge or in-hospital death) will also be recorded.

POTENTIAL RISKS OF INVESTIGATIONAL INTERVENTIONS AND THEIR PREVENTION. Potential risk: Barotrauma. Preventive measures: This potential risk is equally high during CMV or HFO. We also do not anticipate any notable clinical complications due to the use of high-frequency, high mPaw HFO without cuff leak, as its duration of use will not exceed the protocol-pre-specified time limit of 60 min.

POSSIBLE BENEFITS For the participating patient: possible increase in the probability of survival to hospital discharge if HFO-TGI is used as a rescue oxygenation method and detailed TEE evaluation of the cardiac function. For Medical Science: Possible improvement in the understanding of the interaction among ventilatory strategy, heart, and lungs.

ELIGIBILITY:
Inclusion Criteria:

Acute Respiratory Distress Syndrome (ARDS) according to the Berlin Definition Onset of ARDS within the 72 hours preceding study enrollment PaO2/FiO2 of less than 150 mmHg while ventilated with a positive end-expiratory pressure of at least 10 cmH2O Body weight of more than 40 Kg Age 18-75 years

Exclusion Criteria:

Severe air leak (more than one chest tubes per hemithorax with persistent air leak for more than 72 hours) Systolic blood pressure lower than 90 mmHg, despite maximum support with fluids and vasopressor drugs Significant heart disease Severe chronic obstructive pulmonary disease or asthma Intracranial hypertension Chronic interstitial lung disease with bilateral lung infiltrates Lung biopsy or incision during the current admission Previous lung transplantation or bone marrow transplantation Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Right ventricular diastolic area, left ventricular diastolic area as determined by transesophageal echocardiography during the application of the tested ventilatory strategies. | Within 6-7 hours after study enrollment
Eccentricity index as determined by transesophageal echocardiography during the application of the tested ventilatory strategies | Within 6-7 hours after study enrollment

SECONDARY OUTCOMES:
PaO2, PaCO2 and arterial pH during the application of the tested ventilatory strategies | Within 6-7 hours after study enrollment
Mean arterial pressure during the application of the tested ventilatory strategies | Within 6-7 hours after study enrollment
Cardiac index during the application of the tested ventilatory strategies | Within 6-7 hours after study enrollment
Static Compliance of the Respiratory System before and after the application of the tested HFO strategies | Within 6-7 hours after study enrollment

OTHER OUTCOMES:
Occurrence of hypoxemia during the early and intermediate phase of ARDS | Within days 1-10 after study enrollment
Occurrence of in-hospital death and underlying cause(s) | Within days 1-60 after study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Spyros D Mentzelopoulos, MD, PhD, Principal Investigator — University of Athens Medical School, Dept. Intensive Care Medicine; Spyros G Zakynthinos, MD, PhD, Study Chair — University of Athens Medical School, Dept. Intensive Care Medicine
Locations (1):
- Evaggelismos General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ranieri VM, Suter PM, Tortorella C, De Tullio R, Dayer JM, Brienza A, Bruno F, Slutsky AS. Effect of mechanical ventilation on inflammatory mediators in patients with acute respiratory distress syndrome: a randomized controlled trial. JAMA. 1999 Jul 7;282(1):54-61. doi: 10.1001/jama.282.1.54. PMID 10404912
- [Background] Amato MB, Barbas CS, Medeiros DM, Magaldi RB, Schettino GP, Lorenzi-Filho G, Kairalla RA, Deheinzelin D, Munoz C, Oliveira R, Takagaki TY, Carvalho CR. Effect of a protective-ventilation strategy on mortality in the acute respiratory distress syndrome. N Engl J Med. 1998 Feb 5;338(6):347-54. doi: 10.1056/NEJM199802053380602. PMID 9449727
- [Background] Villar J, Kacmarek RM, Perez-Mendez L, Aguirre-Jaime A. A high positive end-expiratory pressure, low tidal volume ventilatory strategy improves outcome in persistent acute respiratory distress syndrome: a randomized, controlled trial. Crit Care Med. 2006 May;34(5):1311-8. doi: 10.1097/01.CCM.0000215598.84885.01. PMID 16557151
- [Background] Ferguson ND, Chiche JD, Kacmarek RM, Hallett DC, Mehta S, Findlay GP, Granton JT, Slutsky AS, Stewart TE. Combining high-frequency oscillatory ventilation and recruitment maneuvers in adults with early acute respiratory distress syndrome: the Treatment with Oscillation and an Open Lung Strategy (TOOLS) Trial pilot study. Crit Care Med. 2005 Mar;33(3):479-86. doi: 10.1097/01.ccm.0000155785.23200.9e. PMID 15753735
- [Background] Fort P, Farmer C, Westerman J, Johannigman J, Beninati W, Dolan S, Derdak S. High-frequency oscillatory ventilation for adult respiratory distress syndrome--a pilot study. Crit Care Med. 1997 Jun;25(6):937-47. doi: 10.1097/00003246-199706000-00008. PMID 9201044
- [Background] Mehta S, Lapinsky SE, Hallett DC, Merker D, Groll RJ, Cooper AB, MacDonald RJ, Stewart TE. Prospective trial of high-frequency oscillation in adults with acute respiratory distress syndrome. Crit Care Med. 2001 Jul;29(7):1360-9. doi: 10.1097/00003246-200107000-00011. PMID 11445688
- [Background] Mentzelopoulos SD, Malachias S, Zintzaras E, Kokkoris S, Zakynthinos E, Makris D, Magira E, Markaki V, Roussos C, Zakynthinos SG. Intermittent recruitment with high-frequency oscillation/tracheal gas insufflation in acute respiratory distress syndrome. Eur Respir J. 2012 Mar;39(3):635-47. doi: 10.1183/09031936.00158810. Epub 2011 Sep 1. PMID 21885390
- [Background] Mentzelopoulos SD, Roussos C, Koutsoukou A, Sourlas S, Malachias S, Lachana A, Zakynthinos SG. Acute effects of combined high-frequency oscillation and tracheal gas insufflation in severe acute respiratory distress syndrome. Crit Care Med. 2007 Jun;35(6):1500-8. doi: 10.1097/01.CCM.0000265738.80832.BE. PMID 17440419
- [Background] Mentzelopoulos SD, Malachias S, Kokkoris S, Roussos C, Zakynthinos SG. Comparison of high-frequency oscillation and tracheal gas insufflation versus standard high-frequency oscillation at two levels of tracheal pressure. Intensive Care Med. 2010 May;36(5):810-6. doi: 10.1007/s00134-010-1822-8. Epub 2010 Mar 16. PMID 20232047
- [Background] Young D, Lamb SE, Shah S, MacKenzie I, Tunnicliffe W, Lall R, Rowan K, Cuthbertson BH; OSCAR Study Group. High-frequency oscillation for acute respiratory distress syndrome. N Engl J Med. 2013 Feb 28;368(9):806-13. doi: 10.1056/NEJMoa1215716. Epub 2013 Jan 22. PMID 23339638
- [Background] Ferguson ND, Cook DJ, Guyatt GH, Mehta S, Hand L, Austin P, Zhou Q, Matte A, Walter SD, Lamontagne F, Granton JT, Arabi YM, Arroliga AC, Stewart TE, Slutsky AS, Meade MO; OSCILLATE Trial Investigators; Canadian Critical Care Trials Group. High-frequency oscillation in early acute respiratory distress syndrome. N Engl J Med. 2013 Feb 28;368(9):795-805. doi: 10.1056/NEJMoa1215554. Epub 2013 Jan 22. PMID 23339639
- [Background] Guervilly C, Forel JM, Hraiech S, Demory D, Allardet-Servent J, Adda M, Barreau-Baumstark K, Castanier M, Papazian L, Roch A. Right ventricular function during high-frequency oscillatory ventilation in adults with acute respiratory distress syndrome. Crit Care Med. 2012 May;40(5):1539-45. doi: 10.1097/CCM.0b013e3182451b4a. PMID 22511135
- [Background] Guervilly C, Roch A, Papazian L. High-frequency oscillation for ARDS. N Engl J Med. 2013 Jun 6;368(23):2233. doi: 10.1056/NEJMc1304344. No abstract available. PMID 23738554
- [Background] Vieillard-Baron A, Price LC, Matthay MA. Acute cor pulmonale in ARDS. Intensive Care Med. 2013 Oct;39(10):1836-8. doi: 10.1007/s00134-013-3045-2. Epub 2013 Aug 2. No abstract available. PMID 23907498
- [Background] Derdak S. High-frequency oscillatory ventilation for acute respiratory distress syndrome in adult patients. Crit Care Med. 2003 Apr;31(4 Suppl):S317-23. doi: 10.1097/01.CCM.0000057910.50618.EB. PMID 12682459
- [Background] Mekontso Dessap A, Charron C, Devaquet J, Aboab J, Jardin F, Brochard L, Vieillard-Baron A. Impact of acute hypercapnia and augmented positive end-expiratory pressure on right ventricle function in severe acute respiratory distress syndrome. Intensive Care Med. 2009 Nov;35(11):1850-8. doi: 10.1007/s00134-009-1569-2. Epub 2009 Aug 4. PMID 19652953
- [Background] Bouferrache K, Vieillard-Baron A. Acute respiratory distress syndrome, mechanical ventilation, and right ventricular function. Curr Opin Crit Care. 2011 Feb;17(1):30-5. doi: 10.1097/MCC.0b013e328342722b. PMID 21157319
- [Background] Ryan T, Petrovic O, Dillon JC, Feigenbaum H, Conley MJ, Armstrong WF. An echocardiographic index for separation of right ventricular volume and pressure overload. J Am Coll Cardiol. 1985 Apr;5(4):918-27. doi: 10.1016/s0735-1097(85)80433-2. PMID 3973294
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Briel M, Meade M, Mercat A, Brower RG, Talmor D, Walter SD, Slutsky AS, Pullenayegum E, Zhou Q, Cook D, Brochard L, Richard JC, Lamontagne F, Bhatnagar N, Stewart TE, Guyatt G. Higher vs lower positive end-expiratory pressure in patients with acute lung injury and acute respiratory distress syndrome: systematic review and meta-analysis. JAMA. 2010 Mar 3;303(9):865-73. doi: 10.1001/jama.2010.218. PMID 20197533
- [Background] Derdak S, Mehta S, Stewart TE, Smith T, Rogers M, Buchman TG, Carlin B, Lowson S, Granton J; Multicenter Oscillatory Ventilation For Acute Respiratory Distress Syndrome Trial (MOAT) Study Investigators. High-frequency oscillatory ventilation for acute respiratory distress syndrome in adults: a randomized, controlled trial. Am J Respir Crit Care Med. 2002 Sep 15;166(6):801-8. doi: 10.1164/rccm.2108052. PMID 12231488
- [Derived] Mentzelopoulos SD, Anninos H, Malachias S, Zakynthinos SG. "Low-" versus "high"-frequency oscillation and right ventricular function in ARDS. A randomized crossover study. J Intensive Care. 2018 Sep 4;6:58. doi: 10.1186/s40560-018-0327-3. eCollection 2018. PMID 30202530